CLINICAL TRIAL: NCT06019481
Title: A Retrospective and Prospective Natural History Study to Examine the Characteristics of Gene-Related Hearing Loss in Pediatric Participants With Biallelic Otoferlin (OTOF) Mutations, Gap Junction Beta 2 (GJB2) Mutations, Or Digenic GJB2/Gap Junction Beta 6 (GJB6) Mutations
Brief Title: A Natural History Study in Pediatric Participants With Hearing Loss Due to OTOF, GJB2, or GJB2/GJB6 Mutations
Acronym: ENSEMBLE
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: DB-100-001
Record Dates: First submitted 2023-08-21; First posted 2023-08-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Congenital Hearing Loss Secondary to Biallelic Mutations in the Otoferlin Gene (OTOF); Biallelic Mutations in the Gap Junction Beta 2 (GJB2) Gene; Digenic Mutations in GJB2/Gap Junction Beta 6 (GJB6) Genes
Keywords: Congenital Hearing Loss; Sensorineural Hearing Loss; Auditory Neuropathy; Pediatric; Cochlear Implant; Otoferlin; GJB2; GJB6; OTOF; Deaf; Hard of hearing; Hearing impaired; Hearing disorder; Fully implantable hearing aid; Child; Infant; ENSEMBLE; Gap Junction Beta 6 Genes; Gap Junction Beta 2 Genes
MeSH Terms: conditions — Hearing Loss, Sensorineural; Auditory neuropathy; Deafness, Autosomal Recessive 9; Hearing Loss; Hearing Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to examine the characteristics of gene-related hearing loss in pediatric participants with biallelic otoferlin (OTOF) Mutations, Gap Junction Beta 2 (GJB2) Mutations, or Digenic GJB2/Gap Junction Beta 6 (GJB6) Mutations. This study will follow the participant for 4 years with annual visits each year.

DETAILED DESCRIPTION:
Former Sponsor Decibel Therapeutics

This is a longitudinal, retrospective and prospective, low interventional study designed to collect data on the natural history of pediatric participants with OTOF, GJB2, or GJB2/GJB6 gene mutations to assess hearing-related outcomes, auditory skills, and speech perception. No investigational product will be administered. At study visits, participants will undergo physiological and behavioral assessments of hearing and vestibular function. Additionally, parents/legal guardians or participants will complete questionnaires that will include the capture of epidemiologic, quality-of-life, auditory and language development, and health resource utilization information.

ELIGIBILITY:
Inclusion Criteria:

* Participant is no older than 7 years (inclusive) at the time of the parent/legal guardian signing the informed consent form (ICF)
* Participant has 1 of the following genotypes and meets the associated audiologic criteria based on physiologic and/or behavioral measures of inner ear function:
* Biallelic pathogenic or likely pathogenic OTOF mutations with severe to profound sensorineural hearing loss (SNHL; ≥ 85 dB HL) and confirmed presence of OAEs
* Biallelic pathogenic and truncating GJB2 mutation(s) with moderate or moderately-severe SNHL (≤41 to <71 dB HL)
* Digenic pathogenic or likely pathogenic mutations in GJB2 and GJB6 genes with mild or worse SNHL (>26 dB HL)
* Participant has at least 1 ear that has not received a cochlear implant (CI)

Exclusion Criteria:

* History of or active participation in an interventional trial related to hearing loss
* History or presence of any other permanent/untreatable hearing loss conditions, including genetic conditions other than those involving biallelic OTOF or GJB2 mutations, or digenic GJB2/GJB6 mutations
* History of treatment with ototoxic drugs

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric participants no older than 7 years, inclusive, who have genetic hearing loss due to OTOF, GJB2, or GJB2/GJB6 mutations.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Hearing-related outcomes | 4 years
  Auditory brainstem response (ABR) intensity
Hearing-related outcomes | 4 years
  Otoacoustic emission (OAEs) amplitudes
Hearing-related outcomes | 4 years
  Pure tone intensity thresholds
Hearing-related outcomes | 4 years
  Speech detection and perception thresholds.

SECONDARY OUTCOMES:
Auditory skills and speech perception over time | 4 years
  Open- and Closed- set Task phoneme accuracy and word comprehension
Auditory skills and speech perception over time | 4 years
  Early Speech Perception (ESP)
Auditory skills and speech perception over time | 4 years
  Pediatric Speech Intelligibility (PSI) test
Auditory skills and speech perception over time | 4 years
  Auditory Skills Checklist (ASC)

OTHER OUTCOMES:
Quality of life over time | 4 years
  Quality of Life-Cochlear Implant (QoL-CI) score
Quality of life over time | 4 years
  Pediatric Quality of Life (PedsQL) Generic Core Scales dimension and total score
Quality of life over time | 4 years
  Hearing Environments and Reflection on Quality of Life (HEAR-QL-26) subscale and overall score

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Patients, Caregivers & Healthcare Providers: Contribute to Genetic Hearing Loss Research — https://portal.sanogenetics.com/study/genetic-hearing-loss-trials